CLINICAL TRIAL: NCT02133482
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 639667 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 639667
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1352.1; 2014-001061-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 639667 (Experimental): single rising doses given as oral solution
  Interventions: Drug: BI 639667
- Placebo (Placebo Comparator): placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo solution
  Arms: Placebo
Drug: BI 639667 — oral solution BI 639667, single rising doses
  Arms: BI 639667

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 639667 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality as well as investigation of linearity and pharmacodynamics (PD) of BI 639667 after single dosing and the assessment of the PK/PD relationship.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. age of 18 to 50 years
3. body mass index (BMI) of 18.5 to 29.9 kg/m2

Exclusion criteria:

1. Any finding in the medical examination (including BP, pulse rate (PR) or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure greater than 140 mmHg, diastolic blood pressure greater than 90 mmHg, or pulse rate outside the range of 50 to 90 mmHg at screening
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with drug-related adverse events | up to 19 days postdose

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 120 hours postdose
Cmax (maximum measured concentration of the analyte in plasma) | up to 120 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim